CLINICAL TRIAL: NCT02529462
Title: Randomised, Controlled, Parallel Clinical Trial on the Efficacy of Pharmacogenetic Information Obtained With NEUROFARMAGEN in the Treatment of Patients With Mental Disorders
Brief Title: Trial to Evaluate Efficacy of Pharmacogenetic Information Obtained With NEUROPHARMAGEN in Treatment of MDD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB-GEN-2013
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2016-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEUROPHARMAGEN-Guided Treatment (Experimental): In the study patient group, the psychiatrist will have the results of the NEUROPHARMAGEN genetic test as supporting information to help him/her select the best treatment for the patient.
  Interventions: Genetic: NEUROPHARMAGEN-Guided Treatment
- Treatment As Usual (Active Comparator): In the control patient group, "treatment as usual" will be selected and prescribed in accordance with routine clinical practice .
  Interventions: Drug: Treatment As Usual

INTERVENTIONS:
Genetic: NEUROPHARMAGEN-Guided Treatment — NEUROPHARMAGEN is a pharmacogenetic test developed by AB-BIOTICS S.A. that enables the specific analysis of Single-Nucleotide Polymorphisms related to the pharmacokinetics and pharmacodynamics of multiple psychoactive drugs. In this arm, psychiatrists have access to the results of the NEUROPHARMAGEN test to support their medication choices
  Other Names: Supportive prescription information from Neuropharmagen test
  Arms: NEUROPHARMAGEN-Guided Treatment
Drug: Treatment As Usual — Clinicians treat psychiatric patients in a naturalistic way, following their routine procedures, without access to the pharmacogenetic information provided by the NEUROPHARMAGEN test
  Other Names: Usual practice
  Arms: Treatment As Usual

SUMMARY:
This study evaluates the efficacy of NEUROPHARMAGEN pharmacogenetic test in the selection of the pharmacological treatments for patients with Major Depressive Disorder (MDD), both with and without psychiatric comorbidities. Patients will be randomly asigned to test-guided treatment prescription or to treatment as usual ina a 1:1 ratio; the results of the test will not be disclosed to the later until the end of the 3-month follow-up period. The study will compare the rate of treatment responders among both groups, based on patient-reported improvement collected by blind telephone interview.

DETAILED DESCRIPTION:
NEUROPHARMAGEN is a genetic test developed by AB-BIOTICS S.A. that enables the specific analysis of Single-Nucleotide Polymorphisms related to the pharmacokinetics and pharmacodynamics of different psychoactive drugs. The aim of the test is to provide the psychiatrist with information that can help him/her identify the most suitable medication for each patient.

In the study group, the psychiatrist will have the results of the NEUROPHARMAGEN test as supporting information to help him/her select the best treatment for the patient. In the control patient group, the treatment will be selected and prescribed in accordance with routine clinical practice.

This is a naturalistic, double-blind, randomized, multicentric clinicaltrial carried out in Spain at psychiatry departments of several public hospitals. The study aims to include a total of 520 patients with MDD, including patient with significant psychiatric comorbidities such as anxiety or substance abuse.

The study will compare groups based on the rate of treatment responders, defined as a score of 2 or less (i.e. "Much better"/"Very much better") in the Patient Global Impression of Improvement scale (PGI-I). This scale will be collected by blind telephone interviewers, so as to have a double-blind assessment (patient and interviewer).

ELIGIBILITY:
Inclusion Criteria at pre-randomization visit:

* Patients with diagnosed for major depressive disorder according to DSM-IV-TR criteria
* Patients who give their written informed consent to participate in the study. In the case of disabled patients, informed consent from the legal representative or responsible relative.
* Patients with a doctor-rated Clinical Global Impression - Severity Scale (CGI-S) score equal to or greater than 4.
* Patients who are diagnosed de novo who, in the doctor's opinion, require medication or are receiving treatment and require an antidepressant, antipsychotic or mood stabiliser as a replacement or additional medication

Exclusion Criteria at pre-randomization visit:

* Patients who, in the investigator's opinion, will not be able to complete the study follow-up.
* Patients who are actively taking part in or who have taken part in another clinical trial in the past 3 months.
* Patients who are pregnant or breast-feeding, or patients who plan to become pregnant within the next 12 months.
* Patients who are or who require treatment with quinidine, cinacalcet and/or terbinafine (potent CYP2D6 inhibitors).

Inclusion criteria at randomization visit:

Patients who meet the screening criteria at the pre-randomisation visit must meet the following criteria at visit 1 to be randomised. Otherwise, they will be excluded from the active follow-up phase. The criteria are:

* Patients with a PGI-I score of 4 or more.
* Patients with a CGI score of 4 or more.
* Patients whose dose of pharmacological treatment, in the doctor's opinion, requires suppression, replacement, addition or modification with an antidepressant, antipsychotic or mood stabiliser.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Sustained response to treatment | 3 months
  The PGI-I scale (Patient Global Impression of Improvement) reports the patient's own assessment of improvement after the therapeutic interventions. It is a single-item questionnaire that assesses the change experienced using a 7-point Likert scale that runs from 1 (very much better) to 7 (very much worse). A sustained response will be considered when the patient reports a PGI-I score of 2 or less, on at least two consecutive assessments, maintained until the end of the follow-up.

SECONDARY OUTCOMES:
Response to treatment | 3 month
  The PGI-I scale (Patient Global Impression of Improvement) reports the patient's own assessment of improvement after the therapeutic interventions. It is a single-item questionnaire that assesses the change experienced using a 7-point Likert scale that runs from 1 (very much better) to 7 (very much worse). A patient will be considered a responder when reporting a PGI-I score of 2 or less (i.e. "much better"/"very much better").
Hamilton Rating Scale for Depression (HAM-D) | 3 months
  HAM-D rates the clinical severity of depression. It has 17 questions, each with three to five possible answers, with scores ranging from 0 to 2 or from 0 to 4, respectively. The total score ranges from 0 to 52 and cut-off scores can be used to classify the depressive disorder.
FIBSER Scale (Frequency, Intensity and Burden of Side Effects Rating) | 3 months
  The scale consists of 3 questions with scores ranging from 0 (no side effects / no impairment) to 6 (intolerable / unable to function / present all of the time).
Clinical Global Impression-Severity scale (CGI-S) | 3 months
  CGI-S is a descriptive scale that provides qualitative information on the severity of the patient's illness. It assesses the severity of the illness using a 7-point Likert scale that runs from 1 (not at all ill) to 7 (among the most extremely ill patients). In this study, both the self-rated (whereby the patient rates his/her own situation) and the doctor-rated versions will be administered so that the doctor can assess the severity of the condition.
Treatment Satisfaction with Medicines Questionnaire (SATMED-Q) | 3 months
  It is a 17-item questionnaire and is a valid scale for any chronic or long-term condition. It is a self-administered questionnaire on treatment satisfaction and it assesses the following areas or dimensions: side effects; effectiveness of the medication; convenience of the medication; impact of the medication on everyday life; medical follow-up of the disease; and the patient's general opinion regarding his/her condition and the medication. All items are assessed using a 5-point Likert scale that runs from "no, not at all" with a value of 0 to "yes, very much" with a value of 4.
Sheehan Disability Inventory (SDI) | 3 months
  SDI is a questionnaire that can be self-administered to measure the disability of patients with mental disorders. It has 3 sub-scales that are scored independently (disability - 3 items, stress - 1 item and perceived social support - 1 item). As each item is scored using a Likert scale from 0 to 10, the maximum possible score is 30.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Menchón, MD, Principal Investigator — Hospital Universitari de Bellvitge; Víctor Pérez, MD, Principal Investigator — Hospital del Mar in Barcelona
Locations (12):
- Spain (12):
  - Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Consorci Sanitari del Maresme, Mataró, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Institut Pere Mata, Reus, Tarragona
  - Hospital Clinic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de Mar, Barcelona
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital 12 de Octubre, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Complejo Hospitalario Universitario de Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menchon JM, Espadaler J, Tuson M, Saiz-Ruiz J, Bobes J, Vieta E, Alvarez E, Perez V. Patient characteristics driving clinical utility in psychiatric pharmacogenetics: a reanalysis from the AB-GEN multicentric trial. J Neural Transm (Vienna). 2019 Jan;126(1):95-99. doi: 10.1007/s00702-018-1879-z. Epub 2018 May 4. PMID 29728861
- [Derived] Perez V, Salavert A, Espadaler J, Tuson M, Saiz-Ruiz J, Saez-Navarro C, Bobes J, Baca-Garcia E, Vieta E, Olivares JM, Rodriguez-Jimenez R, Villagran JM, Gascon J, Canete-Crespillo J, Sole M, Saiz PA, Ibanez A, de Diego-Adelino J; AB-GEN Collaborative Group; Menchon JM. Efficacy of prospective pharmacogenetic testing in the treatment of major depressive disorder: results of a randomized, double-blind clinical trial. BMC Psychiatry. 2017 Jul 14;17(1):250. doi: 10.1186/s12888-017-1412-1. PMID 28705252